CLINICAL TRIAL: NCT01089192
Title: An Open-Label, Randomized, 2-Period, 2-Treatment, Crossover, Single-Dose Bioequivalence Study of Metformin Hydrochloride Extended Release 750 mg Tablets (Test Formulation, Torrent Pharmaceuticals Ltd., India) Versus Glucophage XR® 750 mg Tablet (Reference Formulation, Bristol-Myers Squibb Company, USA) in Healthy Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study of Metformin Hydrochloride Extended Release 750 mg Tablets Versus Glucophage XR® 750 mg Tablet in Healthy Volunteers Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: PK-07-018
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

ARMS (2):
- Torrent's Metformin tablets 750 mg (Experimental)
  Interventions: Drug: Metformin
- Glucophage XR® of Bristol- Myers Squibb Company, USA) (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Objective:

To study Bioequivalence of Metformin Hydrochloride Extended Release 750 mg Tablets (Test formulation, Torrent Pharmaceuticals Ltd., India) Versus Glucophage XR® 750 mg Tablet (Reference formulation, Bristol-Myers Squibb company, USA) in Healthy volunteers under Fasting Conditions.

Study Design:

An Open-Label, Randomized, 2-Period, 2-Treatment, Crossover, Single-Dose Bioequivalence Study

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must meet all of the following criteria in order to be included in the study:

  1. Sex: male.
  2. Age: 18 - 45 years.
  3. Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
  4. Healthy and willing to participate in the study.
  5. Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
  6. Non-smokers or smoker who smokes less than 10 cigarettes a day.

Exclusion Criteria:

* The volunteers will be excluded from the study based on the following criteria:

  1. Clinically relevant abnormalities in the results of the laboratory screening evaluation.
  2. Clinically significant abnormal ECG or Chest X-ray.
  3. Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
  4. Pulse rate less than 50/minute or more than 100/minute.
  5. Oral temperature less than 95°F or more than 98.6°F.
  6. Respiratory rate less than 12/minute or more than 20/minute
  7. Addiction to alcohol or history of any drug abuse within the past 2 years.
  8. Recent History of kidney or liver dysfunction.
  9. History of allergy to the test drug or any drug chemically similar to the drug under investigation.
  10. Administration/ Intake of prescription or OTC medication for two weeks before the study.
  11. Patients suffering from any chronic illness such as arthritis, asthma etc.
  12. HIV, HCV, HBsAg positive volunteers.
  13. Opioids, tetra hydrocannabinoids, amphetamine, barbiturates, benzodiazepine, Cocaine positive volunteers based on urine test.
  14. Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
  15. Administration of any investigational products in the period 0 to 3 months before entry to the study.
  16. Intake of barbiturates or any enzyme-inducing drug in last three months.
  17. History of significant blood loss due to any reason, including blood donation in the past 12 weeks. The total blood loss in last 3 months including for this study will not exceed 350ml.
  18. Existence of any surgical or medical condition, which, in the judgement of the Chief Investigator and/or clinical investigator, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of Volunteers.
  19. Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Torrent Research Centre, Bhat, Gujarat, India

REFERENCES:
- See also: Related Info — http://www.fda.gov/